CLINICAL TRIAL: NCT00934999
Title: A Randomized Comparison of Concomitant Incontinence Procedures Performed With Abdominal Sacral Colpopexy: the Burch Versus Mid-urethral Sling Trial
Brief Title: Comparison of Burch Urethropexy and Mid-urethral Sling Performed Concomitantly With a Sacral Colpopexy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Corewell Health West (Other); Saint Luke's Health System (Other)
Responsible Party: Principal Investigator, Emanuel Trabuco, Assistant Professor, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-007334; 94021001
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Burch (Active Comparator): Patients will receive a Burch urethropexy at the time of an abdominal sacral colpopexy.
  Interventions: Procedure: Burch urethropexy
- Mid-urethral sling (Experimental): Patients will receive a mid-urethral sling at the time of an abdominal sacral colpopexy.
  Interventions: Procedure: Synthetic mid-urethral sling (TVT)

INTERVENTIONS:
Procedure: Burch urethropexy — Patients will undergo a Burch modified Tanagho procedure (in which the anterior vagina is suspended to Cooper's ligament bilaterally using two non-absorbable sutures).
  Arms: Burch
Procedure: Synthetic mid-urethral sling (TVT) — Patients will undergo a polypropylene mid urethral sling as described by the manufacture (Align, Bard Urological, Covington, GA).
  Other Names: TVT
  Arms: Mid-urethral sling

SUMMARY:
I. Specific Aims

Pelvic organ prolapse is a common and distressing condition that is frequently associated with stress urinary incontinence (SUI) and often requires surgical repair. Abdominal sacral colpopexy is the preferred operation for repairing pelvic prolapse. As many as 91% of women with pelvic organ prolapse undergoing sacral colpopexy also experience SUI. In addition, up to 44% of previously continent women develop SUI incontinence after sacral colpopexy: perhaps because a sacral colpopexy may predispose to opening of the bladder neck if secured too tightly. The selection of a surgical procedure to prevent and manage SUI in women undergoing sacral colpopexy is empiric rather than evidence-based. Conceptually, a mid-urethral sling may be more effective than a Burch procedure for preventing urinary leakage because a sling provides outlet resistance beyond the bladder neck and therefore it may compensate for a downward tension on the bladder neck resulting from the sacral colpopexy. Indeed, clinical observations suggest that a mid-urethral sling is effective among women who have persistent urinary incontinence after sacral colpopexy with a Burch procedure. Therefore, the investigators' global hypothesis is that a mid-urethral sling is preferable to a Burch procedure for preventing and improving stress urinary incontinence in women undergoing sacral colpopexy for pelvic organ prolapse. The investigators' SPECIFIC AIMS are to evaluate objective and subjective outcomes at 6, 12 and 24 months in 124 women with urinary incontinence and advanced pelvic organ prolapse. All women will be undergoing a sacral colpopexy and will be randomized to either a Burch procedure or a mid-urethral sling. The primary endpoint is composite continence at 6 months while secondary endpoints will include composite continence and subjective measures of incontinence, patient satisfaction and morbidity associated with these procedures. The investigators' hypotheses are as follows:

1. At 6 months, urinary continence rates will be higher after a mid-urethral than after a Burch procedure. Urine continence will be assessed by composite measure of incontinence: no subjective complaint, no interim treatment, and negative standardized stress test performed by a masked observer. This assessment will be repeated at 12 and 24 months post-operatively to establish the medium term continence of the two procedures. Subjective continence and patient satisfaction measures will be obtained at each of the above visits using standardized questionnaires and pelvic organ support will be quantified by Pelvic Organ Prolapse-Quantification (POP-Q) scores.
2. Early events (e.g., blood loss, operative time, intra-operative complications (vascular, bowel and urological injuries), in-hospital complications (need for transfusion, febrile morbidity, thrombotic events, wound infection, length of stay, duration of bladder catheterization and ileus) and delayed postoperative complications (e.g., wound infection, mesh erosion, bowel obstruction and obstructed voiding) will be collected to compare the safety of each procedure.

ELIGIBILITY:
Inclusion Criteria:

1. older than 21 years of age;
2. with symptomatic pelvic organ prolapse (POP-Q point Aa or C at ≥ -1 cm;
3. who have opted for sacral colpopexy repair of prolapse;
4. who have symptomatic SUI desiring surgical correction or who have occult SUI;
5. who have urethral hypermobility;
6. with a maximal cystometric capacity ≥ 200 cc;
7. who are willing to return for follow-up visit; or
8. who understand and have signed written informed consent to undergo randomization and who has given investigators permission to collect data pertaining to surgical care and follow-up.

Exclusion Criteria:

1. with known or suspected disease that affect bladder function (i.e., multiple sclerosis, Parkinson's Disease, spinal cord injury, etc.);
2. who are pregnant by self report or by positive pregnancy test;
3. who desire to maintain fertility;
4. with history of urethral diverticulum;
5. with a history of radical pelvic surgery or pelvic radiation therapy;
6. who are deemed medically poor candidates for abdominal surgery;
7. Non-ambulatory (including those who ambulate with assistance; or
8. who are actively undergoing chemotherapy or radiation treatment for malignancy.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to compare the proportion of patients who are continent in each group. Continence requires negative standardized stress test performed by a masked observer; no interim re-treatment for SUI; no self reported incontinence (ISI =0) | 6 months

SECONDARY OUTCOMES:
The secondary endpoint is to compare the proportion of patients who have stress specific continence in each group. Stress specific continence requires: fulfilling criteria 1 and 2 above and 3) no self reported SUI specific symptoms. | 6 months
To compared continence, stress specific continence and patient satisfaction between groups at 12 and 24 months. | 12 and 24 months
Compare the safety of the Burch and the mid-urethral sling. | 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel C. Trabuco, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Raju R, Madsen AM, Linder BJ, Occhino JA, Gebhart JB, McGree ME, Weaver AL, Trabuco EC. Defining success after surgical treatment of stress urinary incontinence. Am J Obstet Gynecol. 2024 Aug;231(2):235.e1-235.e16. doi: 10.1016/j.ajog.2024.03.034. Epub 2024 Mar 23. PMID 38527605
- [Derived] Trabuco EC, Linder BJ, Klingele CJ, Blandon RE, Occhino JA, Weaver AL, McGree ME, Gebhart JB. Two-Year Results of Burch Compared With Midurethral Sling With Sacrocolpopexy: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jan;131(1):31-38. doi: 10.1097/AOG.0000000000002415. PMID 29215517